CLINICAL TRIAL: NCT04504318
Title: A Randomized Controlled Trial Comparing Apixaban Versus Enoxaparin Following Microsurgical Breast Reconstruction
Brief Title: Apixaban vs Enoxaparin Following Microsurgical Breast Reconstruction-An RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Arash Momeni, Assistant Professor of Surgery (Plastic Surgery), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-49355
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Tablets; Enoxaparin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban (Experimental): Patients assigned to this group will receive Apixaban 2.5 mg PO BID starting 12 hours after completing skin closure.
  Interventions: Drug: Apixaban 2.5 MG Oral Tablet
- Enoxaparin (Active Comparator): Patients assigned to this group will receive Enoxaparin 40 mg SC QD starting 12 hours after completing skin closure.
  Interventions: Drug: Enoxaparin 40Mg/0.4mL Prefilled Syringe

INTERVENTIONS:
Drug: Apixaban 2.5 MG Oral Tablet — Patients will be assigned to the respective study groups postoperatively upon arrival in the post-anesthesia care unit. Hence, surgeons are blinded at the time of surgery as to study group assignment. Chemoprophylaxis will continue for the duration of the hospitalization.
  Arms: Apixaban
Drug: Enoxaparin 40Mg/0.4mL Prefilled Syringe — Patients will be assigned to the respective study groups postoperatively upon arrival in the post-anesthesia care unit. Hence, surgeons are blinded at the time of surgery as to study group assignment. Chemoprophylaxis will continue for the duration of the hospitalization.
  Arms: Enoxaparin

SUMMARY:
Subcutaneous enoxaparin is currently the gold standard for VTE chemoprophylaxis. However, the efficacy of chemoprophylaxis with subcutaneous enoxaparin is affected by patient-level factors, thus, resulting in VTE events despite guideline-compliant prophylaxis. A population at particular risk is the growing number of patients who undergo autologous breast reconstruction. Direct oral anticoagulants (DOAC) might be a less invasive, yet, more efficacious mode of chemoprophylaxis in this patient population. Hence, the proposed work has the potential to cause a paradigm shift in chemoprophylaxis guidelines in a large population of patients undergoing plastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) women
* Scheduled to undergo unilateral or bilateral microsurgical breast reconstruction with free abdominal flaps (i.e. muscle-sparing transverse rectus abdominis musculocutaneous [TRAM] and/or deep inferior epigastric artery perforator [DIEP]) flap)
* Caprini score of 6 or greater.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Contraindication to the use of apixaban or enoxaparin
* Active bleeding
* History of bleeding disorder
* History of coagulopathy
* History of heparin-induced thrombocytopenia
* History of liver disease
* History of renal disease (creatinine clearance <30 mL/min; serum creatinine >1.6 mg/dL)
* Major neurosurgical intervention (brain/spine) within the past 90 days
* Ophthalmologic procedure within the past 90 days
* Uncontrolled hypertension
* History of alcohol and/or substance abuse
* Need for therapeutic anticoagulation
* Pregnant or Nursing

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Momeni, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 82 participants signed informed consent; 76 were allocated to treatment.
Period: Overall Study
Arm/Group | Apixaban | Enoxaparin
Started | 37 | 39
Completed | 37 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Enoxaparin | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10) | 53 (11) | 53 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 76
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 39 | 76

OUTCOME MEASURES:

1. Primary Outcome: Apixaban vs. Enoxaparin - Number of Participants With Bleeding Events
Description: To examine the rate of bleeding events in patients receiving oral apixaban versus subcutaneous enoxaparin following microsurgical breast reconstruction
Time Frame: 90-day events
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Enoxaparin
Number analyzed (Participants) | 37 | 39
Participants | 1 | 1

2. Secondary Outcome: Apixaban vs. Enoxaparin - Number of Participants With Venous Thromboembolism (VTE) Events
Description: To examine the rate of VTE events in patients receiving oral apixaban versus subcutaneous enoxaparin following microsurgical breast reconstruction
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Enoxaparin
Number analyzed (Participants) | 37 | 39
Participants | 6 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 90 days from the surgery date.
Arm/Group | Apixaban | Enoxaparin
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/37 | 1/39
Other Adverse Events (participants affected / at risk) | 6/37 | 5/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=37) | Enoxaparin (N=39)
Bleeding Event (Surgical and medical procedures) | 1 (1) | 1 (1) — Subject had bleeding event prior to administration of medication
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=37) | Enoxaparin (N=39)
Cellulitis at donor site (abdomen) (Surgical and medical procedures) | 1 (1) | 1 (1)
Wound dehsicence at breast (Surgical and medical procedures) | 1 (1) | 1 (1)
Breast Cellulitis (Surgical and medical procedures) | 1 (1) | 1 (1)
Mastectomy skin necrosis (Surgical and medical procedures) | 1 (1) | 1 (1)
Wound deshiscence at abdomen (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Surgical and medical procedures) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT04504318/Prot_SAP_000.pdf